CLINICAL TRIAL: NCT01347151
Title: A Comparison of Cervical Spine Movement During Tracheal Intubation Using the Pentax or the Glidescope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Assistant Professor Nalinee Kovitwanawong, Department of anesthesiology Faculty of Medicine Prince of Songkla University Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Glide VS Pentax
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: C-spine Movement During Intubation
Keywords: Glide scope; Pentax; C spine movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glide scope (Experimental)
  Interventions: Device: The glidescope video laryngoscopy
- Pentax airway scope (Experimental)
  Interventions: Device: The Pentax airwayscope

INTERVENTIONS:
Device: The glidescope video laryngoscopy
  Arms: Glide scope
Device: The Pentax airwayscope
  Other Names: The Pentax airwayscope (Pentax AWS; Pentax, Tokyo, Japan)
  Arms: Pentax airway scope

SUMMARY:
Both Glide scope and Pentax laryngoscope are video laryngoscope that provide the better view with minimal cervical spine movement. This study wants to compare cervical spine movement during intubation when using these two devices. The C-spine motion will be recorded by using fluoroscopic video to measure the angular displacement of the vertebrae.

DETAILED DESCRIPTION:
The primary outcome is the angular displacement of the vertebrae and secondary outcome is the hemodynamic changes after intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-75 years old
* Elective noncardiac surgery requiring general anesthesia with tracheal intubation

Exclusion Criteria:

* Gastroesophageal reflux disease
* Body mass index greater than 35 kg/m2
* Possibility of pregnancy
* Previous neck surgery
* Unstable C-spine/ C-spine abnormality
* Known difficult airway
* Suspected difficult airway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
the angular displacement of the vertebrae | 30 seconds
  during intubation

SECONDARY OUTCOMES:
the hemodynamic changes after intubation. | 15 minutes
  after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Nalinee Kovitwanawong, MD, Principal Investigator — Depatment of Anesthesiology Faculty of Medicine Prince of Songkla University Thailand
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand